CLINICAL TRIAL: NCT04396665
Title: Feasibility of an Educational Intervention for the Prevention of Breast Cancer by Modifying Risk Behaviors Through a Web Application
Brief Title: Breast Cancer: Feasibility of an Educational Intervention
Acronym: PRECAM-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oviedo (Other)
Responsible Party: Principal Investigator, Rubén Martín Payo, Principal Investigator, University of Oviedo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 147/19
Record Dates: First submitted 2020-03-29; First posted 2020-05-20 (Actual); Results first posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Women's Health: Neoplasm of Breast
Keywords: Breast neoplasm; Health Promotion; Dietary; Phycical activity; Breast cancer risk
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Precam Group (Intervention Group) (Experimental): 150 Women without breast cancer, aged from 25 to 50 years old
  Interventions: Behavioral: Precam
- Control Group (No Intervention): 150 Women without breast cancer, aged from 25 to 50 years old

INTERVENTIONS:
Behavioral: Precam — 6 months Web-App intervention related with: diet, physical activity, self-care and breast cacner risk prevention
  Arms: Precam Group (Intervention Group)

SUMMARY:
Aim: To evaluate the viability of an educational intervention for the prevention of breast cancer risk and the modification of their risk behaviors through the use of a web application in women living in the Principality of Asturias.

Design: pilot test Population: 300 women without breast cancer living in Asturias. 25 to 50 years old. Informed consent signed.

Variables: personal characteristics (age, status, educational level, occupation), MIC index, dietary characteristics, level of physical activity, presence of known risks of breast cancer (number of children, breastfeeding, oral contraceptives, family history of cancer, previous cancer, breast density and knowledge related with breast cancer prevention.

Intervention:

* Intervention Group:6 months intervention using a web-app related with personal care and breast cancer risks, diet and physical activity.
* Control Group: no intervention.

DETAILED DESCRIPTION:
Aim: To evaluate the viability of an educational intervention for the prevention of breast cancer risk and the modification of their risk behaviors through the use of a web application in women living in the Principality of Asturias.

Design: pilot test Population: 300 women without breast cancer living in Asturias. 25 to 50 years old. They are recluted for a previous study developed by the same research team. An information document and a written consent was given for the women. Those who signed the consent are included.

The randomization for intervention or control group are doing based on the where the city where the women home is located. the objective of this distribution is to avoid contact between women from different groups.

Variables: personal characteristics (age, status, educational level, civil status), MIC index, dietary characteristics, level of physical activity, knowledge related with breast cancer symptoms and risk factors.

Intervention:

The 6 months intervention are going to be developed using a web-app. The intervention is based on the Behavior Change Wheel model. Capacity and motivation are going to be the determinants on which it will work using for it interventions based on education, persuasion and modeling among others.

Intervention Group: 6 months intervention using a web-app related. The web-app includes some sections:

* Information related with breast cancer risk.
* Breast self examination. Written text and videos done by a nurse.
* Physical exercise. Written text and videos done by a physiotherapist .
* Dietary information. Written text and videos done by a nutrition expert.

The Control Group are not going to receive intervention during the study period time. After that, women are going to be access to the web-app.

Statistical analysis

Descriptive statistics will be carried out (means, standard deviation, CI and percentages). In addition, at the end of the study, in order to determine the factibility of the educational intervention, the variation of the intra-group data (from pre to psot-test) and between the groups in post-test will be compared using the chi-square test. , t-student or Mann-Whitney U, for qualitative or quantitative data respectively.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed
* Capability to use internet

Exclusion Criteria:

* Breast cancer diagnosis duting the intervention

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 224 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Martin Payo, PhD, Principal Investigator — University of Oviedo
Locations (1):
- University of Oviedo, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: No
Anonymizes data are going to be published but we are not going to analizase individual data.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Precam Group (Intervention Group) | Control Group
Started | 134 | 90
Completed | 99 | 83
Not Completed | 35 | 7

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group: Women in the Intervention group
- Control Group: Women in the Control group
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 134 | 90 | 224
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (6.685) | 38.2 (7.334) | 39.5 (7.017)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134 | 90 | 224
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 134 | 90 | 224
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Spain | 134 | 90 | 224
Studies [Count of Participants; unit: Participants]
  Non universitary | 51 | 24 | 75
  University | 83 | 66 | 149
Civil status [Count of Participants; unit: Participants]
  Single | 39 | 36 | 75
  Married or similar | 79 | 46 | 125
  Divorced or widowed | 16 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of an Educational Intervention: Adherence to the Intervention
Description: Participants that finish the intervention
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 134 | 90
Participants | 99 | 83

2. Primary Outcome: Feasibility of an Educational Intervention: Drop Out After the Intervention Period
Description: People that did not finish the intervention
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: Women in the intervention group
- Control: Women in the control group
Arm/Group | Intervention | Control
Number analyzed (Participants) | 134 | 90
Participants | 35 | 7

3. Primary Outcome: Number of Diet and Activity Recommendations
Description: Mean number of recommendations done by the participants
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Number of recommendations
Groups:
- Intervention Group: 150 Women without breast cancer, aged from 25 to 50 years old
  Precam: 6 months Web-App intervention related with: diet, physical activity, self-care and breast cacner risk prevention
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 99 | 83
Number of recommendations | 9.38 (1.789) | 8.28 (2.265)

4. Primary Outcome: Breast Cancer Awareness
Description: Using 2 dimensions of MARA questionnaire (Scale title)1) knowledge of risk factors of breast cancer (range 0=worst score to 9=better score); 2) knowledge of signs and symptoms of breast cancer (range 0=worst score to 9=better score)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 99 | 83
units on a scale
  Risk factors knowledge | 2.04 (1.531) | 1.31 (1.239)
  Symptoms knowledge | 3.61 (0.636) | 3.38 (0.809)

ADVERSE EVENTS:
Description: Adverse Events were not monitored/assesed
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-09): https://cdn.clinicaltrials.gov/large-docs/65/NCT04396665/Prot_SAP_000.pdf